CLINICAL TRIAL: NCT00129584
Title: Endobronchial Valve for Emphysema Palliation Trial (VENT)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Emphasys Medical (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 630-0001
Record Dates: First submitted 2005-08-10; First posted 2005-08-12 (Estimated); Last update posted 2009-08-18 (Estimated); Status verified 2009-08

CONDITIONS: Chronic Obstructive Pulmonary Disease; Emphysema
Keywords: Endobronchial Valve (EBV) Procedure; Bronchoscopic Lung Volume Reduction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Emphysema; Epstein-Barr Virus Infections

INTERVENTIONS:
Procedure: Emphasys Endobronchial Valve and procedure

SUMMARY:
The purpose of this study is to assess the safety and efficacy of the Emphasys Endobronchial Valve (EBV) and procedure (with pulmonary rehabilitation) compared to optimal medical management (with pulmonary rehabilitation) in patients with heterogeneous emphysema.

DETAILED DESCRIPTION:
Background:

Emphysema, caused primarily by smoking, is characterized by the gradual, irreversible breakdown of tissue and loss of elastic recoil within the lungs, causing them to lose the ability to expel air and efficiently absorb oxygen. As this chronic condition inexorably progresses, the diseased, hyperinflated areas of the lung eventually fill the chest cavity, leaving less and less volume available for the viable lung tissue.

Lung volume reduction surgery (LVRS) has been shown to offer relief to patients suffering from emphysema when other treatment options fail. Researchers have continued to refine both technique and patient selection in order to improve outcomes. The objective of lung volume reduction is to eliminate dysfunctional, over-inflated regions of lung. Results similar to surgical removal have been obtained by plication (folding) and stapling without tissue removal. These results suggest that isolation of the dysfunctional lung region can achieve similar results to tissue removal.

The paradoxical effect of improving lung function by removing (or isolating) lung tissue demonstrates that breathlessness due to emphysema is a function of mechanical inefficiencies in addition to loss of gas-transfer surface area and other physiological mechanisms. At least in some patients, the mechanical compromise is the primary cause of their pulmonary incapacitation and these patients can benefit by addressing their inability to effectively inhale and exhale. Because LVRS reduces trapped gas, others have speculated that results similar to LVRS could be achieved bronchoscopically by reducing the volume of the hyperinflated regions with, or without, atelectasis.

Emphasys has developed a bronchoscopic approach to block inspiratory airflow into targeted, hyperinflated regions of the lung, while permitting exhaled gas to escape. This approach may lead to lung volume reduction and provide some of the clinical benefits of LVRS without the high risks and costs associated with such an invasive surgical procedure.

Comparison:

The primary object of this study is to assess the safety and efficacy of the Emphasys Endobronchial Valve (EBV) and procedure (with pulmonary rehabilitation) compared to medical management (with pulmonary rehabilitation) in patients with heterogeneous emphysema.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed by high-resolution computed tomography (HRCT) with eligible heterogeneous disease distribution
* Forced expiratory volume in 1 second (FEV1) < 45% predicted
* Total lung capacity (TLC) > 100% predicted
* Residual volume (RV) > 150% predicted
* Post rehabilitation 6 minute walk test > 140m
* Non-smoking for 4 months

Exclusion Criteria:

* Prior lung transplant, LVRS, median sternotomy, bullectomy or lobectomy
* History of recurrent respiratory infections
* Evidence of large bullae (>30% of either lung) in a non-target lobe
* FEV1 < 15% predicted
* Diffusing capacity for carbon monoxide (DLCO) < 20% predicted

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Start 2004-01

PRIMARY OUTCOMES:
Pulmonary function testing at various time points through one year
Exercise tolerance at various time points through one year
Major complications at various time points through one year

SECONDARY OUTCOMES:
Pulmonary function testing at various time points through one year
Quality of life measures at various time points through one year
Other adverse event rates at various time points through one year

CONTACTS AND LOCATIONS:
Overall Officials: Frank C Sciurba, MD, Principal Investigator — University of Pittsburgh Medical Center

REFERENCES:
- [Background] Celli BR, Cote CG, Marin JM, Casanova C, Montes de Oca M, Mendez RA, Pinto Plata V, Cabral HJ. The body-mass index, airflow obstruction, dyspnea, and exercise capacity index in chronic obstructive pulmonary disease. N Engl J Med. 2004 Mar 4;350(10):1005-12. doi: 10.1056/NEJMoa021322. PMID 14999112
- [Background] Sciurba FC, Rogers RM, Keenan RJ, Slivka WA, Gorcsan J 3rd, Ferson PF, Holbert JM, Brown ML, Landreneau RJ. Improvement in pulmonary function and elastic recoil after lung-reduction surgery for diffuse emphysema. N Engl J Med. 1996 Apr 25;334(17):1095-9. doi: 10.1056/NEJM199604253341704. PMID 8598868
- [Background] Martinez FJ, de Oca MM, Whyte RI, Stetz J, Gay SE, Celli BR. Lung-volume reduction improves dyspnea, dynamic hyperinflation, and respiratory muscle function. Am J Respir Crit Care Med. 1997 Jun;155(6):1984-90. doi: 10.1164/ajrccm.155.6.9196106.
- [Background] Sabanathan A, Sabanathan S, Shah R, Richardson J. Lung volume reduction surgery for emphysema. A review. J Cardiovasc Surg (Torino). 1998 Apr;39(2):237-43. PMID 9639013
- [Background] Geddes D, Davies M, Koyama H, Hansell D, Pastorino U, Pepper J, Agent P, Cullinan P, MacNeill SJ, Goldstraw P. Effect of lung-volume-reduction surgery in patients with severe emphysema. N Engl J Med. 2000 Jul 27;343(4):239-45. doi: 10.1056/NEJM200007273430402. PMID 10911005
- [Background] Gelb AF, McKenna RJ Jr, Brenner M, Schein MJ, Zamel N, Fischel R. Lung function 4 years after lung volume reduction surgery for emphysema. Chest. 1999 Dec;116(6):1608-15. doi: 10.1378/chest.116.6.1608. PMID 10593784
- [Background] Gierada DS, Yusen RD, Villanueva IA, Pilgram TK, Slone RM, Lefrak SS, Cooper JD. Patient selection for lung volume reduction surgery: An objective model based on prior clinical decisions and quantitative CT analysis. Chest. 2000 Apr;117(4):991-8. doi: 10.1378/chest.117.4.991. PMID 10767229
- [Background] Russi EW, Bloch KE, Weder W. Functional and morphological heterogeneity of emphysema and its implication for selection of patients for lung volume reduction surgery. Eur Respir J. 1999 Jul;14(1):230-6. doi: 10.1034/j.1399-3003.1999.14a39.x. PMID 10489857
- [Background] Rogers RM, Coxson HO, Sciurba FC, Keenan RJ, Whittall KP, Hogg JC. Preoperative severity of emphysema predictive of improvement after lung volume reduction surgery: use of CT morphometry. Chest. 2000 Nov;118(5):1240-7. doi: 10.1378/chest.118.5.1240. PMID 11083670
- [Background] Gelb AF, Zamel N, McKenna RJ Jr, Brenner M. Mechanism of short-term improvement in lung function after emphysema resection. Am J Respir Crit Care Med. 1996 Oct;154(4 Pt 1):945-51. doi: 10.1164/ajrccm.154.4.8887590.
- [Background] Swanson SJ, Mentzer SJ, DeCamp MM Jr, Bueno R, Richards WG, Ingenito EP, Reilly JJ, Sugarbaker DJ. No-cut thoracoscopic lung plication: a new technique for lung volume reduction surgery. J Am Coll Surg. 1997 Jul;185(1):25-32. doi: 10.1016/s1072-7515(97)00021-5. PMID 9208957
- [Background] Hoppin FG Jr. Theoretical basis for improvement following reduction pneumoplasty in emphysema. Am J Respir Crit Care Med. 1997 Feb;155(2):520-5. doi: 10.1164/ajrccm.155.2.9032188.
- [Background] Iwasaki M, Nishiumi N, Kaga K, Kanazawa M, Kuwahira I, Inoue H. Application of the fold plication method for unilateral lung volume reduction in pulmonary emphysema. Ann Thorac Surg. 1999 Mar;67(3):815-7. doi: 10.1016/s0003-4975(98)01302-2. PMID 10215234
- [Background] Kuwahira I, Iwasaki M, Kaga K, Iwamoto T, Tazaki G, Ishii M, Inoue H, Ohta Y. Effectiveness of the fold plication method in lung volume reduction surgery. Intern Med. 2000 May;39(5):381-4. doi: 10.2169/internalmedicine.39.381. PMID 10830177
- [Background] Fishman A, Martinez F, Naunheim K, Piantadosi S, Wise R, Ries A, Weinmann G, Wood DE; National Emphysema Treatment Trial Research Group. A randomized trial comparing lung-volume-reduction surgery with medical therapy for severe emphysema. N Engl J Med. 2003 May 22;348(21):2059-73. doi: 10.1056/NEJMoa030287. Epub 2003 May 20. PMID 12759479
- [Background] Toma TP, Hopkinson NS, Hillier J, Hansell DM, Morgan C, Goldstraw PG, Polkey MI, Geddes DM. Bronchoscopic volume reduction with valve implants in patients with severe emphysema. Lancet. 2003 Mar 15;361(9361):931-3. doi: 10.1016/S0140-6736(03)12762-6. PMID 12648974
- [Derived] Valipour A, Herth FJ, Burghuber OC, Criner G, Vergnon JM, Goldin J, Sciurba F, Ernst A; VENT Study Group. Target lobe volume reduction and COPD outcome measures after endobronchial valve therapy. Eur Respir J. 2014 Feb;43(2):387-96. doi: 10.1183/09031936.00133012. Epub 2013 Jul 11. PMID 23845721
- [Derived] Herth FJ, Noppen M, Valipour A, Leroy S, Vergnon JM, Ficker JH, Egan JJ, Gasparini S, Agusti C, Holmes-Higgin D, Ernst A; International VENT Study Group. Efficacy predictors of lung volume reduction with Zephyr valves in a European cohort. Eur Respir J. 2012 Jun;39(6):1334-42. doi: 10.1183/09031936.00161611. Epub 2012 Jan 26. PMID 22282552
- [Derived] Sciurba FC, Ernst A, Herth FJ, Strange C, Criner GJ, Marquette CH, Kovitz KL, Chiacchierini RP, Goldin J, McLennan G; VENT Study Research Group. A randomized study of endobronchial valves for advanced emphysema. N Engl J Med. 2010 Sep 23;363(13):1233-44. doi: 10.1056/NEJMoa0900928. PMID 20860505
- [Derived] Strange C, Herth FJ, Kovitz KL, McLennan G, Ernst A, Goldin J, Noppen M, Criner GJ, Sciurba FC; VENT Study Group. Design of the Endobronchial Valve for Emphysema Palliation Trial (VENT): a non-surgical method of lung volume reduction. BMC Pulm Med. 2007 Jul 3;7:10. doi: 10.1186/1471-2466-7-10. PMID 17711594